CLINICAL TRIAL: NCT06842446
Title: Evaluating a New Diagnostic Strategy for Suspected DVT Consisting of Point of Care D-dimer, AI-based Prediction Model and Compression Ultrasound
Brief Title: Systematic Machine Learning Algorithm for Rapid Thrombosis Detection
Acronym: DVT-SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 682139
Record Dates: First submitted 2024-12-04; First posted 2025-02-24 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Machine Learning; POC D-dimer; POC Ultrasound
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- All participants (Experimental): All participants will be treated the same way.
  Interventions: Diagnostic Test: POC D-dimer; Diagnostic Test: POC ultrasound; Diagnostic Test: Machine learning model

INTERVENTIONS:
Diagnostic Test: POC D-dimer — POC D-dimer will be compared to laboratory D-dimer in hospital setting and used in a machine learning model
Diagnostic Test: POC ultrasound — Point of care (POC) ultrasound performed by ED physicians compared to ultrasound performed by radiologist. POC ultrasound 3 point examination performed by ED physician will be compared with POC ultrasound full leg examination performed by ED physician.
Diagnostic Test: Machine learning model — The DSS will be compared to the usual strategy. It will also be estimated how many participants where DVT could have been excluded without ultrasound.
  Other Names: Decision support system

SUMMARY:
The goal of this clinical trial is to compare the use of a machine learning-based algorithm and point-of-care D-dimer to laboratory D-dimer and compression ultrasound to exclude deep vein thrombosis in the under extremities in patients referred to a medical department suspected of having deep vein thrombosis. The main aim is to answer are if a machine learning algorithm and point of care D-dimer can exclude deep vein thrombosis in more patients than clinical assessment and D-dimer alone.

DETAILED DESCRIPTION:
All participants will follow the usual diagnostic algorithm used for patients with suspected DVT referred to Ostfold Hospital (all patients are examined by a physician, D-dimer is analyzed in all patients, ultrasound is performed by a radiologist in patients with positive D-dimer). In addition to usual care, POC D-dimer, POC ultrasound (performed by ED physicians), blood sampling for biobanking, and photographies of the under extremities will be performed. The machine learning model will be tested to see if the prediction is correct. In participants where ultrasound is performed, it will also be assessed whether the machine learning algorithm could have excluded the participant without the use of ultrasound. None of the additional procedures will have any impact on the patient diagnostics or treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the ED due to suspicion of DVT
* Age ≥ 18 years
* Able to give informed consent

Exclusion Criteria:

* Ongoing use of anticoagulation for more than 72 hours
* Previous participation in the study
* Life expectancy of less than three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-01-05 (Estimated); Study Completion 2029-01-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the new strategy (POC D-dimer, ML-based prediction model, POC CUS by emergency physician) | From enrollment to the end of the primary assessment period (90 days)
  Evaluate the safety of a new strategy consisting of POC D-dimer and an ML-based prediction model followed by CUS performed by emergency physicians by comparing the new strategy's safety with our standard care by measuring the proportion of patients in whom DVT is excluded according to the new strategy but was diagnosed with DVT by standard care or in whom DVT is diagnosed within the 90-day follow up.

SECONDARY OUTCOMES:
Evaluate the efficiency of the new strategy | From enrollment to the end of the primary assessment period (90 days)
  The proportion of patients in whom DVT can be ruled out by the ML-based prediction model with POC D-dimer compared to the efficiency of Wells score and laboratory D-dimer
Validate the safety and efficiency of the ML-based prediction model | From enrollment to the end of the primary assessment period (90 days)
  Safety will be determined by the proportion of patients in whom DVT is excluded by the ML-model but diagnosed by standard care. Efficiency will be determined by the proportion of patients in whom DVT can be excluded by the ML-based model
Evaluate concordance between CUS performed by emergency physicians and radiologists. | From time of enrollment until time of ultrasound examination performed by radiologist, assessed up to 48 hours.
  Determine the proportion of false negative and false positive diagnosis of DVT in emergency physician-performed ultrasound compared with ultrasound performed by radiologists.
Evaluate concordance between POC D-dimers in an ED setting and laboratory D-dimers. | From enrollment to the completion of D-dimer analysis, assessed up to 24 hours.
  Compare the two POC D-dimers with the STA-Liatest D-dimer and Siemens INNOVANCE by direct comparison of the true/false positive/negative results.
Evaluate the hypothetical time to be completed for the novel strategy compared to the standard strategy. | From time of enrollment until time of discharge from the emergency department either discharged from the hospital or hospitalized, assessed up to 24 hours.
  Estimating the total management time defined as time from ED registration to ED discharge in patients evaluated according to the new strategy compared to standard care.
Evaluate the safety of a limited ultrasound protocol (two-point and proximal) compared to full-leg CUS performed by emergency physicians and radiologists | 90 days after enrollment.
  Estimating the proportion of patients in whom DVT was ruled out by the limited ultrasound protocol but was diagnosed with DVT by the whole-leg ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- Østfold Hospital Trust, Sarpsborg, Norway

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share IPD with other researchers are not yet decided because it has not yet been discussed.